CLINICAL TRIAL: NCT03271099
Title: Patient Navigation as Part of the Cancer Survivorship Care Plan at a Safety Net Institution
Brief Title: Patient Navigation in Cancer Survivorship at a Safety Net Institution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-36781
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Cancer
Keywords: survivorship; navigation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care
- Navigator (Experimental): Patient navigator services provided as part of survivorship care plan
  Interventions: Other: Navigator

INTERVENTIONS:
Other: Navigator — Patient Navigation services will be provided to try to eliminate barriers in pursuing survivorship surveillance
  Other Names: navigation
  Arms: Navigator

SUMMARY:
This study seeks to enroll patients receiving a Survivorship Care Plan following curative therapy for cancer. Participants will be randomly assigned to receive usual care or to be followed by a Patient Navigator as part of their Survivorship Care Plan.

DETAILED DESCRIPTION:
This study seeks to enroll patients receiving a Survivorship Care Plan following curative therapy for cancer. Participants will be randomly assigned to receive usual care or to be followed by a Patient Navigator as part of their Survivorship Care Plan.

Study participation for all participants will be for up to 9 months, with study visits approximately every 3 months, based on standard clinical follow-up. All participants will be administered quality of life surveys by a Clinical Research Associate at study entry, mid-study (approximately 3-6 months) and at study completion.

The following factors will be compared between arms:

* Missed/kept appointments
* Use of urgent/emergent care
* Quality of Life in relation to survivorship care
* Participants lost to care

ELIGIBILITY:
Inclusion Criteria:

* Stage I, II, III or IVa Cancer diagnosis (may include Solitary plasmacytoma, Diffuse Large B-Cell Lymphoma (DLBCL), ductal carcinoma in situ (DCIS) of the breast)
* Completed treatment with curative intent within the past 12 months. (May be on maintenance therapy.)

Exclusion Criteria:

* Distant Metastatic disease
* Non-curable disease
* Recurrence of disease prior to enrollment
* Require ongoing navigation from the treatment navigator
* Enrolled/active in another randomized study (Project SUPPORT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Missed appointments | 9 months
  The research team will document the number of cancer care appointments scheduled and of those, how many appointments were missed (obtained by medical record and by patient report in case a visit was outside of study institution).

SECONDARY OUTCOMES:
Urgent/emergent care | 9 months
  The research team will document the number of urgent/emergent care visits attended within the study period of 9 months (obtained by medical record and by patient report in case a visit was outside of study institution).
Cancer Needs Distress | 9 months
  Participants will rate their feelings about 39 specific cancer needs on a 5 point scale from "Not a Problem" to "Very Severe Problem" using the Cancer Needs Distress Inventory (CaNDI) tool. Total scores can range from 39 to 195. Lower scores are associated with less cancer related distress.
New Survivor Survey | 9 months
  Participants will rate their understanding about 16 specific aspects of survivorship care on a 4 point scale from "Strongly Disagree" to "Strongly Agree" using the Preparing for Life as a New Survivor (PLANS) Scale. Total scores can range from 16 to 48. Lower scores are associated with less understanding of the survivorship care process.
Lost to Care | 9 months
  The research team will document the number of participants lost to care, based on consecutive missed cancer care visits.

CONTACTS AND LOCATIONS:
Overall Officials: Minh Tam Truong, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No